CLINICAL TRIAL: NCT02750202
Title: Prophylactic Vaccines as Therapy: Prevention of Recurrence of Extensive Genital Warts
Brief Title: Effectiveness Study of Human Papilloma Virus (HPV) Vaccines to Prevent Recurrence of Genital Warts
Acronym: TheraVACCS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pretoria (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Professor Greta Dreyer, Professor, University of Pretoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Merck-MISP-53183
Record Dates: First submitted 2016-04-12; First posted 2016-04-25 (Estimated); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Genital Warts
Keywords: Genital warts; HPV types; HPV vaccine; Cervical cytology; Therapeutic vaccine; Quadrivalent HPV vaccine
MeSH Terms: conditions — Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadrivalent HPV vaccine (Active Comparator): Three doses of 4 HPV vaccine is given at registered intervals.
  Interventions: Biological: Quadrivalent HPV vaccine
- Hepatitis B vaccine (Sham Comparator): Three doses of Hepatitis B vaccine is given at the same intervals as the quadrivalent HPV vaccine.
  Interventions: Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: Quadrivalent HPV vaccine — Quadrivalent HPV vaccine doses administered intramuscular as 3 separate 0.5 ml doses at month 0, month 2 and month 6.
  Other Names: Gardasil; 4 HPV vaccine; q HPV vaccine
  Arms: Quadrivalent HPV vaccine
Biological: Hepatitis B vaccine — Hepatitis B vaccine doses administered intramuscular as 3 separate 0.5 ml doses at month 0, month 2 and month 6.
  Other Names: Hep B vaccine
  Arms: Hepatitis B vaccine

SUMMARY:
Large genital warts are frequently diagnosed in general gynaecology and oncology clinics in South Africa. Medical and destructive therapy for small warts is generally very effective, however unique problems posed by large or extensive genital warts are not so easily solved and treatment of affected patients remains very challenging. Recurrences are common especially among immune-compromised women. This study will test whether giving the quadrivalent human papilloma virus (HPV) vaccine to women with extensive genital warts prior to surgical treatment will improve outcomes. Investigators hypothesize that pre-treatment with HPV vaccine can play a role in the control of both malignant and benign HPV disease in women with and without HIV infection through stimulation of the antibody response. In addition, HPV types and other associated diseases will be studied in women receiving HPV vaccine and placebo.

DETAILED DESCRIPTION:
Patient selection:

Female patients referred or presenting with genital warts at each site will be eligible and evaluated against the inclusion and exclusion criteria.

Women who are clinically or severely immune-compromised will not be included into the study, but both HIV negative and HIV infected women will be included. Seventy-five women with large or recurrent genital warts will be recruited for this study from 2 sites in South Africa.

Recruitment:

Women with genital warts will be evaluated for inclusion into the study. Those who fit the inclusion criteria and are without any of the exclusion criteria will be fully informed and invited to participate. The first target will be to recruit the first seventy-five consecutive eligible patients who have signed written consent; recruitment for the study will be done for at least 24 months.

First clinical visit:

* Evaluation genital lesions:

On study entry tumour size and position will be documented graphically and photographically and viral typing from the vulva wart and cervix will be done using Roche Linear Array test.

* Evaluation immune status:

HIV status and CD 4/CD 8 count will be recorded and tested and the serum will be collected for antibody testing. Cervical disease of clinical significance will be excluded or treatment offered if relevant.

* Randomization:

Patients will be randomized to receive either quadrivalent HPV or Hepatitis B vaccine.

* Vaccination:

The participants assigned to the test group will be administered quadrivalent HPV vaccine in three doses as recommended by the manufacturer. Participants assigned to the control group will receive Hepatitis B vaccine in three doses as recommended by the manufacturer.

Follow-up clinical visits: week 8, week 16 and week 24:

* Evaluation genital lesions:

Three follow up visits will be scheduled two months apart at which time the lesion size will be recorded.

* Evaluation immune status:

After month 6 or the third visit, the serum will again be collected for antibody level testing.

* Treatment decision:

According to the clinical response as measured at month six and onwards, locally destructive or surgical treatment will be allowed according to the preference of the clinician and as determined by clinical factors.

Follow up after treatment:

* Follow up will be done at six monthly intervals.
* Evaluation genital lesions:

At these visits lesion size will be determined and documented. HPV typing on the cervical and vulval lesions will be repeated at least once.

* Further treatment of warts:

If needed, repeat surgery and/or local destruction will be allowed and documented. These will be around week 48 and week 72, or study exit

Study exit:

* Participants will exit the study in week 72.
* In the absence of harm as determined at interim analysis or suggested by participant disease history, researchers will be unblinded for participant status at study exit and alternative vaccines will be offered to each of these women.

ELIGIBILITY:
Inclusion Criteria:

* Female patient > 16 years
* Presence of vulvo vaginal genital warts: largest tumour diameter > 3 cm OR Tumour on labia minora and labia majora OR bilateral > 1 cm each side OR Tumour in vagina/cervix as well as on vulva > 1 cm lesion each
* HIV negative or HIV infected and CD4 ≥ 300 cells/mm3 OR viral load controlled OR anti retro-viral (ARV) compliant > 6 months

Exclusion Criteria:

* Pregnant of planned pregnancy within 6 months
* Not able to comprehend study method or not able to attend all study visits
* Previous HPV vaccination
* Active known opportunistic infection or malignancy including Pneumocystis pneumonia (PCP),Pulmonary tuberculosis (PTB), oesophageal Candida or Kaposi sarcoma or lymphoma
* Known allergy to vaccines or content of vaccine
* Previous radiation for genital warts

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greta G Dreyer, MMed(O&G)PhD, Principal Investigator — University of Pretoria
Locations (2):
- South Africa (2):
  - Steve Biko Academic Hospital, Pretoria, Gauteng
  - Tygerberg Hospital, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on referral at two academic medical centers in South Africa between July 2018 and June 2021. First participant was enrolled on 20 July 2018 and the last participant was enrolled in June 2021
Pre-assignment Details: A total of 52 participants met the inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine
Started | 28 | 24
Completed | 25 | 23
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (9.96) | 32.9 (10.27) | 35.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 52
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Self-reported tobacco smoking [Count of Participants; unit: Participants] | 2 | 5 | 7
Self-reported medical diseases [Count of Participants; unit: Participants] | 7 | 10 | 17
HIV-positivity [Count of Participants; unit: Participants] | 25 | 21 | 46
White cell count [Mean (Standard Deviation); unit: cells x 10^9/l] | 6.1 (1.95) | 6.8 (2.38) | 6.4 (2.18)
Haemoglobin [Mean (Standard Deviation); unit: g/dl] | 11.7 (1.58) | 12.1 (1.31) | 11.9 (1.48)
Platelet count [Mean (Standard Deviation); unit: cells x 10^9 /l] | 323 (99.2) | 331 (73.0) | 327 (88.4)
Alkaline phosphatase (blood test) [Mean (Standard Deviation); unit: U/l] | 94 (21.1) | 88 (26.5) | 91 (23.9)
Alanine transaminase (blood test) [Mean (Standard Deviation); unit: U/l] | 23 (14.6) | 20 (7.8) | 21 (12.0)
Bilirubin total [Mean (Standard Deviation); unit: µmol/l] | 6.5 (4.2) | 6.1 (4.4) | 6.3 (4.3)
Total protein (blood test) [Mean (Standard Deviation); unit: g/l] | 79 (6.6) | 80 (6.9) | 79 (6.7)
Serum sodium [Mean (Standard Deviation); unit: mmol/l] | 138 (1.9) | 138 (2.6) | 138 (2.3)
Serum potassium [Mean (Standard Deviation); unit: mmol/l] | 4.4 (0.77) | 4.4 (0.95) | 4.4 (0.86)
Serum chloride [Mean (Standard Deviation); unit: mmol/l] | 106 (2.3) | 105 (2.9) | 106 (2.6)
Total serum carbon dioxide [Mean (Standard Deviation); unit: mmol/l] | 22 (2.1) | 23 (3.6) | 23 (2.9)
Serum urea [Mean (Standard Deviation); unit: mmol/l] | 3.2 (0.8) | 3.7 (1.5) | 3.4 (1.2)
Number of vulva lesions [Count of Participants; unit: Participants]
  1-5 lesions | 7 | 5 | 12
  6-10 lesions | 6 | 7 | 13
  11-15 lesions | 7 | 3 | 10
  15+ lesions | 8 | 9 | 17
Diameter of largest vulva lesion [Mean (Standard Deviation); unit: mm] | 61 (62) | 81 (184) | 70 (133)
Number of cervico-vaginal lesions (per category) [Count of Participants; unit: Participants]
  No visible lesion | 10 | 12 | 22
  1-5 lesions | 14 | 6 | 20
  6-10 lesions | 1 | 1 | 2
  11-15 lesions | 0 | 3 | 3
  15+ lesions | 3 | 2 | 5
Diameter of largest cervico-vaginal lesion - estimated [Mean (Standard Deviation); unit: mm] | 15 (10) | 12 (8) | 14 (9)
Cytology results (baseline) [Count of Participants; unit: Participants]
  Normal | 9 | 5 | 14
  Atypical Squamous Cells of Undetermined Significance (ASCUS) [slightly abnormal] | 0 | 2 | 2
  Low-Grade Squamous Intraepithelial Lesion (LSIL) [monitor for progression] | 9 | 7 | 16
  High-Grade Squamous Intraepithelial Lesion (HSIL) [needs treatment] | 10 | 10 | 20
Cervix HPV prevalence [Count of Participants; unit: Participants]
  High-risk HPV positive | 23 | 16 | 39
  Low-risk HPV positive | 24 | 19 | 43
Vulvar HPV prevalence (baseline) [Count of Participants; unit: Participants]
  High-risk HPV positive | 18 | 17 | 35
  Low-risk HPV positive | 25 | 21 | 46
Cervical histopathology (LLETZ biopsies) [Count of Participants; unit: Participants] — Population: Not all participants required LLETZ treatment
  Participants
    Normal: number analyzed (Participants) | 8 | 9 | 17
    Normal | 0 | 2 | 2
    Cervical Intraepithelial Neoplasia Grade 2 (CIN2) [moderately abnormal cells, needs treatment]: number analyzed (Participants) | 8 | 9 | 17
    Cervical Intraepithelial Neoplasia Grade 2 (CIN2) [moderately abnormal cells, needs treatment] | 0 | 4 | 4
    Cervical Intraepithelial Neoplasia Grade 3 (CIN3) [severely abnormal cells, needs treatment]: number analyzed (Participants) | 8 | 9 | 17
    Cervical Intraepithelial Neoplasia Grade 3 (CIN3) [severely abnormal cells, needs treatment] | 8 | 3 | 11
Vulvar histopathology [Count of Participants; unit: Participants]
  Condylomata acuminata (genital warts - benign, better outcome) | 14 | 12 | 26
  Vulvar Intraepithelial Neoplasia Grade 1 (VIN1, better outcome) [needs monitoring] | 2 | 1 | 3
  Vulvar Intraepithelial Neoplasia grade 2 (VIN2, worse outcome) [needs treatment] | 0 | 2 | 2
  Vulvar Intraepithelial Neoplasia 3 (VIN3, worse outcome) [needs treatment] | 10 | 8 | 18
  Vulvar squamous cell carcinoma (worst outcome) [needs treatment] | 4 | 1 | 5
Treatment type for vulvar lesions [Count of Participants; unit: Participants]
  Surgery and or cautery | 19 | 20 | 39
  Cryotherapy | 1 | 2 | 3
  Surgery followed by imiquimod | 1 | 0 | 1
  Imiquimod only | 3 | 2 | 5
  No treatment during trial | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in the Maximum Size of the Genital Wart Lesion Over the Trial Period (as Measured in mm)
Description: The number of participants in whom the size of the genital wart lesion(s) measured smaller at Week8, Week24 and Week60 as compared to their baseline measurement (all measured in mm).
Time Frame: Baseline, week 8, 24, 60
Population: Some participants were lost to follow up after Week 28
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine
Number analyzed (Participants) | 28 | 24
Participants
  Week0 vs Week8 | 8 | 6
  Week0 vs Week24 | 11 | 7
  Week0 vs Week60: number analyzed (Participants) | 23 | 22
  Week0 vs Week60 | 19 | 22

2. Secondary Outcome: Number of Participants Who Acquire Measurable Levels of HPV Type Specific Antibodies During the First 18 Months of the Trail as Measured Using a Competitive Luminex Immuno-assay (cLIA; Reported in Milli-Merck Units [mMU]/ml)
Time Frame: Week 36+
Reporting Status: Not Posted, anticipated posting 2028-02

3. Secondary Outcome: Number of Participants Who Change From HPV 6 DNA Positive in Warts to Negative at Week 72
Description: The number of participants who change from HPV 6 DNA positive in warts to HPV 6 DNA negative at week 72
Time Frame: Baseline, week 72
Population: Only participants who were positive for HPV6 at baseline were assessed for possible conversion to HPV6-negative at Week 72
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine
Number analyzed (Participants) | 20 | 21
Participants
  Number of participants HPV6 positive at W0 (wart lesion) | 10 | 9
  Number of participants who changed from HPV6 positive at W0 to HPV6 negative at Week72 (wart lesion): number analyzed (Participants) | 10 | 9
  Number of participants who changed from HPV6 positive at W0 to HPV6 negative at Week72 (wart lesion) | 1 | 2

4. Secondary Outcome: Number of Participants Who Change From HPV 11 DNA Positive in Warts to Negative at Week 72
Description: The number of participants who change from HPV 11 DNA positive in warts to negative at week 72
Time Frame: Baseline, week 72
Population: Only participants who were positive for HPV11 at baseline were assessed for possible conversion to HPV11-negative at Week 72
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine
Number analyzed (Participants) | 20 | 21
Participants
  Number of participants HPV11 positive at W0 (wart lesion) | 7 | 11
  Number of participants who changed from HPV11 positive at W0 to HPV11 negative at W72 (wart lesion): number analyzed (Participants) | 7 | 11
  Number of participants who changed from HPV11 positive at W0 to HPV11 negative at W72 (wart lesion) | 1 | 2

5. Secondary Outcome: Number of Participants Who Change From HPV 16 DNA Positive at Baseline to Negative at Week 60
Description: The number of participants who change from HPV 16 DNA positive at baseline to negative at week 60
Time Frame: Baseline, week 60
Population: Only participants who were positive for HPV16 at baseline were assessed for possible conversion to HPV16-negative at Week 60
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine
Number analyzed (Participants) | 20 | 21
Participants
  Number of participants HPV16 positive at W0 (wart lesion) | 8 | 7
  Number of participants who changed from HPV16 positive at W0 to HPV16 negative at W60 (wart lesion): number analyzed (Participants) | 8 | 7
  Number of participants who changed from HPV16 positive at W0 to HPV16 negative at W60 (wart lesion) | 2 | 1

6. Secondary Outcome: Number of Participants Who Change From HPV 18 DNA Positive at Baseline to Negative at Week 60
Description: The number of participants who change from HPV 18 DNA positive at baseline to negative at week 60
Time Frame: Baseline, week 60
Population: Only participants who were positive for HPV18 at baseline were assessed for possible conversion to HPV18-negative at Week 60
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine
Number analyzed (Participants) | 20 | 21
Participants
  Number of participants HPV18 positive at W0 (wart lesion) | 3 | 2
  Number of participants who changed from HPV18 positive at W0 to HPV18 negative at W60 (wart lesion): number analyzed (Participants) | 3 | 2
  Number of participants who changed from HPV18 positive at W0 to HPV18 negative at W60 (wart lesion) | 0 | 2

7. Other Pre Specified Outcome: Number of Participants Who Change From HIV Negative at Baseline to Positive at Week 48
Description: The number of participants who change from HIV negative at baseline to positive at week 48
Time Frame: Baseline, week 48
Population: Number of participants who change from HIV negative at baseline to positive at week 48. Only HIV-negative participants were assessed at Week 48.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine
Number analyzed (Participants) | 28 | 24
Participants
  Number of participants who were HIV-negative at baseline | 3 | 3
  The number of participants who changed from HIV negative at baseline to HIV-positive at week 48: number analyzed (Participants) | 3 | 3
  The number of participants who changed from HIV negative at baseline to HIV-positive at week 48 | 0 | 0

8. Other Pre Specified Outcome: Number of Participants Who Require Surgical Treatment of Warts at Any of the Clinical Assessments During the Trial, as Judged by the Attending Clinician.
Description: The number of participants who require surgical treatment of warts at any of the clinical assessments during the trial, as judged by the attending clinician.
Time Frame: Week 24, 72
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine
Number analyzed (Participants) | 28 | 24
Participants
  Require surgical treatment of warts at W28 | 21 | 18
  Require surgical treatment of warts at W72 | 2 | 1

9. Other Pre Specified Outcome: Number of Participants Who Require Surgical Treatment of Cervical Disease at Any of the Clinical Assessments During the Trial, as Judged by the Attending Clinician.
Description: The number of participants who require surgical treatment of cervical disease at any of the clinical assessments during the trial, as judged by the attending clinician.
Time Frame: Week 24, 72
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine
Number analyzed (Participants) | 28 | 24
Participants
  Need Large Loop Excision of the Transformation Zone (LLETZ) at Week24 | 10 | 10
  Need Large Loop Excision of the Transformation Zone (LLETZ) at Week72 | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 year after Week0 (first vaccine dose administrated)
Arm/Group | Quadrivalent HPV Vaccine | Hepatitis B Vaccine
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/24
Other Adverse Events (participants affected / at risk) | 0/28 | 0/24

LIMITATIONS AND CAVEATS:
COVID-19 disruptions impacted hugely on this study: gynaecologic outpatient-, HIV- and other clinics scaled down/closed down, and because these clinics were our main sources in recruiting patients, we experienced a huge challenge to find patients fulfilling our inclusion criteria. Participants also experienced financial stress or lost jobs & subsequently moved to family homes in rural areas, that led to a number of our participants LTFU. We had to adapt, modify or delay our research project.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT02750202/Prot_ICF_000.pdf